CLINICAL TRIAL: NCT03859739
Title: A Single-Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Anti-Retroviral Activity of MK-8558 Monotherapy in Anti-Retroviral-Naïve HIV-1 Infected Participants
Brief Title: Safety, Tolerability, Pharmacokinetics, and Anti-Retroviral Activity of MK-8558 Monotherapy in Anti-Retroviral-Naïve HIV-1 Infected Participants (MK-8558-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8558-002; MK-8558-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Panel A. MK-8558 400 mg (Experimental): Single oral dose of MK-8558 administered at 400 mg following a 10-hour fast.
  Interventions: Drug: MK-8558
- Panel B. MK-8558 at dose level 2 (Experimental): Single oral dose of MK-8558 administered at dose level 2 following a 10-hour fast. Dose level 2 shall not exceed 900 mg. Per protocol, dose will be selected following review of data from panel A.
  Interventions: Drug: MK-8558
- Panel C. MK-8558 at dose level 3 (Experimental): Single oral dose of MK-8558 administered at dose level 3 following a 10-hour fast. Dose level 3 shall not exceed 1600 mg. Per protocol, dose will be selected following review of data from panel B.
  Interventions: Drug: MK-8558
- Panel D. MK-8558 at dose level 4 (Experimental): Single oral dose of MK-8558 administered at dose level 4 following a low-fat breakfast. Dose level 4 shall not exceed 1600 mg. Per protocol, Panel D is optional pending results of Panels A-C, and dose will be selected following review of data from panel C.
  Interventions: Drug: MK-8558

INTERVENTIONS:
Drug: MK-8558 — Single dose of MK-8558 administered as a tablet at a dose up to 1600 mg.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and anti-retroviral activity of MK-8558 monotherapy in anti-retroviral-naïve human immunodeficiency virus type 1 (HIV-1) infected participants. The primary hypothesis is that at a dose that exhibits an acceptable safety and tolerability profile, MK-8558 has superior anti-retroviral activity compared to historical placebo data.

ELIGIBILITY:
Inclusion Criteria:

* Other than having HIV infection, is in good health based on medical history, physical examination, vital sign (VS) measurements, and laboratory safety tests, at the pre-study (screening) visit and/or prior to administration of the study drug
* Is documented as being HIV-1 positive
* Has a screening plasma HIV-1 ribonucleic acid (RNA) ≥ 2,500 copies/mL within 30 days prior to the treatment phase of this study
* Has a screening plasma cluster of differentiation 4+ (CD4+) T-cell count of >200/mm^3
* Is antiretroviral therapy (ART)-naïve
* Is willing to receive no other ART prior to Day 11 post-dose of the trial, unless the physician/Investigator believes that there is a strong indication to start ART before Day 11
* Has a Body Mass Index (BMI) ≤35 kg/m^2
* Males must agree to abstinence, or barrier contraception plus partner contraception, unless confirmed to be azoospermic due to vasectomy or medical cause, for at least 35 days after the last dose of MK-8558
* Females must not be pregnant or breastfeeding, and must be a woman of nonchildbearing potential, or a woman of childbearing potential using highly effective birth control with low user dependency or who is abstinent on a long-term and persistent basis during the intervention period and at least 35 days after the last dose of study medication

Exclusion Criteria:

* Has acute (primary) HIV-1 infection
* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic (with the exception of Gilbert's disease), immunological (outside of HIV-1 infection), renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated or has a history of a clinically significant psychiatric disorder (with the exception of situational depression) of the last 5 years
* Has a history of cancer unless disease is adequately treated and deemed "cured"
* Has an estimated creatinine clearance (CrCl) ≤ 90 mL/min
* Has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food, or has hereditary galactose intolerance, lactase deficiency, or glucose-galactose malabsorption
* Is positive for hepatitis B surface antigen
* Has a history of chronic hepatitis C unless there has been documented cure
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-study (screening) visit
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study, until the post-study visit. There may be certain medications that are permitted
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the pre-study (screening) visit. The window will be derived from the date of the last visit in the previous study
* Is under the age of legal consent or not capable of giving consent
* Has been committed to an institution by way of official or judicial order
* Is an excessive smoker (i.e., more than 10 cigarettes/day) and is unwilling to restrict smoking to ≤10 cigarettes per day
* Consumes more than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day. Participants who consume 4 glasses of alcoholic beverages per day may be enrolled at the discretion of the investigator
* Consumes excessive amounts, defined as more than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Has a positive urine drug screen (except for cannabis) at screening and/or pre-dose; rechecks are allowed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Charite Research Organisation GmbH ( Site 0001), Berlin, Germany
- Matei Bals Infectious Diseases Institute ( Site 0002), Bucharest, București, Romania

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Human Immunodeficiency Virus Type 1 (HIV-1) infection, who were naïve to anti-retroviral therapy (ART) between 18 and 60 years old (inclusive) were enrolled in this study.
Groups:
- MK-8558 400 mg: Single oral dose of MK-8558 administered at 400 mg following a 10-hour fast.
- MK-8558 900 mg: Single oral dose of MK-8558 administered at 900 mg following a 10-hour fast.
- MK-8558 1600 mg: Single oral dose of MK-8558 administered at 1600 mg following a 10-hour fast.
- MK-8558 900 mg Low-Fat: Single oral dose of MK-8558 administered at 900 mg following a low-fat meal.
Period: Overall Study
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Started | 5 | 6 | 6 | 4
Completed | 5 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat | Total
Number analyzed (Participants) | 5 | 6 | 6 | 4 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.2 (5.0) | 39.3 (12.6) | 32.5 (9.8) | 32.3 (18.6) | 33.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 5 | 6 | 6 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 6 | 4 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 5 | 5 | 4 | 19
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma HIV-1 Ribonucleic Acid (RNA) Concentration
Description: Plasma was collected at baseline and at 168 hours post-dose to determine the change from baseline in HIV-1 ribonucleic acid (RNA) concentration. The log10 plasma HIV-RNA was measured and analyzed based on a longitudinal data analysis (LDA) model containing fixed effects for dose level and time.
Time Frame: Baseline and 168 hours post-dose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. One participant from the 900 mg treatment group was excluded from analysis due to important protocol deviation.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
log10 copies/mL | -0.82 [-1.42 to -0.21] | -1.00 [-1.61 to -0.39] | -1.61 [-2.16 to -1.06] | -1.81 [-2.48 to -1.13]
Statistical Analysis 1: Comparison: MK-8558 400 mg; It was hypothesized that the true mean difference in the plasma HIV-1 RNA reduction from baseline between MK-8558 and placebo is ≥ 1.4 log10 copies/mL; Test type: Superiority — Adjusted by Placebo data pooled from historical placebo data from recent monotherapy studies in HIV-1 infected participants (NCT00100048, NCT01466985, NCT01152255, and NCT01353898) and fitted with a LDA model containing fixed effects for study and time, and a random effect for participants; Posterior Mean Difference = -0.79 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8558 and placebo ≤ -1.4 copies/mL was 2.44 %
Statistical Analysis 2: Comparison: MK-8558 900 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Posterior Mean Difference = -0.97 — PP of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8558 and placebo ≤ -1.4 copies/mL was 7.60%
Statistical Analysis 3: Comparison: MK-8558 1600 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Posterior Mean Difference = -1.58 — PP of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8558 and placebo ≤ -1.4 copies/mL was 74.99%
Statistical Analysis 4: Comparison: MK-8558 900 mg Low-Fat; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Posterior Mean Difference = -1.78 — PP of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8558 and placebo ≤ -1.4 copies/mL was 87.41%

2. Primary Outcome: Number of Participants Experiencing ≥1 Adverse Event (AE)
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to 35 days post-dose
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 6 | 6 | 4
Participants | 4 | 3 | 4 | 0

3. Primary Outcome: Number of Participants Who Discontinued From the Study Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to 35 days post-dose
Population: All participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 6 | 6 | 4
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to 168 Hours (AUC0-168) for MK-8558 in Plasma
Description: Plasma was collected from pre-dose up to 168 hours post-dose in order to determine the AUC0-168 for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μM
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
hr*μM | 1740 (24.2) | 2780 (20.7) | 5740 (36.3) | 5340 (15.6)

5. Secondary Outcome: Area Under the Concentration-Time Curve From 0 up to the Last Quantifiable Time-Point (AUC0-last) for MK-8558 in Plasma
Description: Plasma was collected from pre-dose up to 504 hours post-dose in order to determine the AUC0-last for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μM
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
hr*μM | 2650 (32.9) | 4450 (16.2) | 9680 (42.6) | 8580 (9.6)

6. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to Infinity (AUC0-inf) for MK-8558 in Plasma
Description: Plasma was collected from pre-dose up to 504 hours post-dose in order to determine the AUC0-inf for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μM
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
hr*μM | 2840 (37.3) | 4870 (14.7) | 11100 (48.9) | 9520 (9.8)

7. Secondary Outcome: Maximum Observed Concentration (Cmax) for MK-8558 in Plasma
Description: Plasma was collected from pre-dose up to 504 hours post-dose in order to determine the Cmax for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
μM | 24.3 (21.7) | 36.7 (28.9) | 77.2 (28.9) | 72.6 (14.3)

8. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) for MK-8558 in Plasma
Description: Plasma was collected from pre-dose up to 504 hours post-dose in order to determine the Tmax for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
Hours | 4.00 [1.50 to 4.00] | 4.00 [4.00 to 5.00] | 4.50 [4.00 to 8.02] | 4.02 [4.00 to 5.00]

9. Secondary Outcome: Concentration at 168 Hours Post-Dose (C168hr) for MK-8558 in Plasma
Description: Plasma was collected at 168 hours post-dose in order to determine the C168hr for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
μM | 5.59 (44.0) | 9.55 (17.7) | 20.5 (43.4) | 18.8 (8.1)
Statistical Analysis 1: Comparison: MK-8558 400 mg; The posterior probability (PP) that the true GM C168hr is ≥ 9.0 μM was calculated using a non-informative (Jeffrey's) prior under an assumption of normality of log C168hr; Test type: Other; Standard Error (SE) = 0.146 — PP that the true C168hr in plasma MK-8558 is ≥ 9.0 μM was 0.25%
Statistical Analysis 2: Comparison: MK-8558 900 mg; The PP that the true GM C168hr is ≥ 9.0 μM was calculated using a non-informative (Jeffrey's) prior under an assumption of normality of log C168hr; Test type: Other; SE = 0.146 — PP that the true C168hr in plasma MK-8558 is ≥ 9.0 μM was 65.41%
Statistical Analysis 3: Comparison: MK-8558 1600 mg; [analysis description as in outcome 9, analysis 2]; Test type: Other; SE = 0.133 — PP that the true C168hr in plasma MK-8558 is ≥ 9.0 μM was 99.99%
Statistical Analysis 4: Comparison: MK-8558 900 mg Low-Fat; [analysis description as in outcome 9, analysis 2]; Test type: Other; SE = 0.163 — PP that the true C168hr in plasma MK-8558 is ≥ 9.0 μM was 99.98%

10. Secondary Outcome: Apparent Clearance (CL/F) for MK-8558
Description: Plasma was collected from pre-dose up to 504 hours post-dose in order to determine the CL/F for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
L/hr | 0.315 (37.3) | 0.412 (14.7) | 0.321 (48.9) | 0.211 (9.8)

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for MK-8558
Description: Plasma was collected from pre-dose up to 504 hours post-dose in order to determine the Vz/F for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
Liters | 56.6 (21.9) | 84.4 (27.5) | 79.9 (30.8) | 45.6 (20.5)

12. Secondary Outcome: Terminal Half Life (t1/2) for MK-8558
Description: Plasma was collected from pre-dose up to 504 hours post-dose in order to determine the t1/2 for MK-8558. Data were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
Number analyzed (Participants) | 5 | 5 | 6 | 4
Hours | 125 (24.9) | 142 (20.1) | 173 (22.7) | 150 (20.6)

ADVERSE EVENTS:
Time Frame: Adverse events: Up to 35 days post-dose; All-cause mortality: Up to 9 weeks after randomization.
Description: All participants who received at least one dose of treatment.
Arm/Group | MK-8558 400 mg | MK-8558 900 mg | MK-8558 1600 mg | MK-8558 900 mg Low-Fat
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/6 | 1/6 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 3/6 | 4/6 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8558 400 mg (N=5) | MK-8558 900 mg (N=6) | MK-8558 1600 mg (N=6) | MK-8558 900 mg Low-Fat (N=4)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8558 400 mg (N=5) | MK-8558 900 mg (N=6) | MK-8558 1600 mg (N=6) | MK-8558 900 mg Low-Fat (N=4)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT03859739/Prot_SAP_000.pdf